CLINICAL TRIAL: NCT07192380
Title: Shift Hours' Impact on Fatigue and Tracking of Eye Dynamics
Acronym: SHIFTED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IMADIS Technologies et Services (Industry)
Collaborators: Lyon Neuroscience Research Center (CRNL) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PSI-24-05; ID-RCB (Registry Identifier: 2024-A02843-44)
Record Dates: First submitted 2025-09-05; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Sleep Deprivation; Sleepiness; Eye-Tracking Technology; Radiologists; Tomography; Electroencephalography
Keywords: Night-Shift; Radiology; performance; Eye-tracking; Fatigue; Eye strain
MeSH Terms: conditions — Sleep Deprivation; Sleepiness; Fatigue; Asthenopia | interventions — Electroencephalography; Actigraphy; Eye-Tracking Technology; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Experimental): Radiologists taking measurements after a night shift and after a night's rest
  Interventions: Device: Electroencephalogram; Device: Actigraphy; Device: Eye Tracking; Other: Questionnaires

INTERVENTIONS:
Device: Electroencephalogram — EEG measurement to assess attentional state
  Other Names: EEG
Device: Actigraphy — Evaluation of sleep-wake phases 24 hours prior to eye tracking measurement
  Other Names: Actimetry
Device: Eye Tracking — Assessment of ocular parameters during controlled eye tracking: guided saccade task followed by analysis of chest scans to detect pulmonary embolism. Measurement of ocular saccade parameters (distance, velocity), fixation time and pupil diameter.
  Measurements performed twice: after a night on call and after a night of rest.
  Other Names: Oculometry
Other: Questionnaires — Measurements of sleepiness (Karolinska Sleep Scale KSS, Epworth Sleep Scale ESS), mental fatigue (EVA Scale), insomnia (Insomnia Severity Index, ISI) and chronotype (Morningness Eveningness Questionnaire, MEQ)
  * Inclusion visit: MEQ
  * Before the first evaluation: ISI, KSS, ESS, EVA
  * Before the second evaluation: ISI, KSS, ESS, EVA

SUMMARY:
The goal of this clinical trial is to learn how night shift-induced sleep debt affects oculomotor patterns, attentional state, and diagnostic performance in emergency radiologists.

The main questions it aims to answer are:

* Does sleep debt from a night shift alter oculomotor parameters, as eyes movements (speed and amplitude), fixation duration, pupil size?
* Does a night shift impact radiologists' diagnostic accuracy, attentional state, and perceived fatigue? Researchers will compare radiologists after a night shift (sleep-deprived) with the same radiologists after a night of rest (control) to see if fatigue-related changes affect both visual exploration strategies and diagnostic performance.

Participants will:

* Perform a guided saccade task assessed by eye tracking (primary endpoint),
* Read thoracic CT scans (with and without pulmonary embolism cases) to assess diagnostic performance and visual exploration patterns,
* Undergo EEG recording to measure attentional state,
* Complete self-report questionnaires on sleepiness and fatigue.

DETAILED DESCRIPTION:
Rationale Physician burnout is a significant problem, particularly for emergency physicians and radiologists working in emergency imaging. Over the past 15 years, the workload of 'emergency radiologists' has increased significantly, impacting their job satisfaction and perceived health. Night shifts and reduced recovery time disrupt the sleep-wake cycle, leading to decreased cognitive performance and increased stress. Fatigue at work is closely linked to a higher risk of medical errors. Radiologists face high demands on attention, pressure to report quickly, and the need to interpret complex images, all of which contribute to errors.

Eye tracking has been used to analyze radiologists' visual search patterns, However, few studies have examined the impact of work patterns, particularly night shifts, on these behaviors. It is important to study the effect of night shift fatigue on radiologists' eye movement patterns and cognitive abilities, and to relate these findings to their diagnostic performance.

Research Hypothesis The investigators hypothesize that eye movement patterns and attention during medical image reading will be influenced by sleep debt and ocular fatigue induced by night shifts.

The investigators therefore aim to compare radiologists' eye movement patterns during medical image reading, as measured by oculometry, and their attentional state, as measured by EEG, according to their sleep debt within the IMADIS Group.

STUDY DESIGN Study type Longitudinal (non-randomized controlled trial design), single-center, multi-site study (IMADIS Group)

Study procedure Inclusion Before any research-related act or intervention, the investigator will inform the participant and obtain their free, informed, and written consent to take part in the study.

Each participant will perform 2 measures. Radiologists will undergo each measurement in an order determined by their work schedule within the IMADIS Group (after on-call night or after night of rest).

Measure After the participant's consent is obtained, data will be collected using the case report form, including demographic data and sleep-related information. This visit will also serve to schedule all other study visits with the participant.

Actimeters (Geneactive) will be handed over to participants with instructions for use (continuous wear during the day and night preceding each measurement). The actimeter is worn day and night before the oculometry measurement to record their sleep-wake rhythms.

A chronotype questionnaire will also be administered. Morningness-Eveningness Questionnaire (MEQ, ordinal 16-86) Eye -tracking and EEG measurements Upon arrival at the IMADIS Group on-call center (between 08:00 and 10:00 after a night of rest) or before leaving the center after an on-call night (between 08:00 and 10:00), participants will complete brief questionnaires (Mental Fatigue VAS score, Karolinska Sleepiness Scale (KSS, ordinal 0-9), Insomnia Severity Index (ISI, ordinal 0-28), and Epworth Sleepiness Scale (ESS, ordinal 0-14).) while being fitted with the EEG headset. This will be followed by an eye tracker calibration phase.

The eye-tracking study scenario will then be launched on the Tobii Pro Lab platform. It will include a guided saccade task of approximately 5 minutes, followed by an observation phase comprising 10 videos simulating navigation through multiple slices of a thoracic CT scan. The videos will differ between measurement phases but equivalent.

During the experimentation, recording of the brain activity modulations and attentional state (Theta, Alpha, Beta, Gamma waves) will be performed with EPOC X EEG headset (EMOTIV).

Statistical aspects Required sample size For this study, the investigators will use a significant change in the slope of the relationship between peak saccadic velocity and saccadic amplitude. Based on the results of prvious studies and considering two comparison groups with an effect size of 0.8, the required sample size is 8 participants to achieve a statistical power of at least 80% with a 5% type I error risk.

The calculations were performed using the power.anova.test function from the stat package (R software®, version 4.0.5). The investigators chose to add 32 participants to account for potential missing or poor-quality data, leading to a total of 40 participants. This estimate is supported by the literature..

Statistical methods Univariate descriptive analyses Descriptive analyses will be performed on quantitative and ordinal variables. Data will be summarised for the entire sample and separately by group, reporting frequencies and percentages for qualitative variables, and means, medians, standard deviations, and quartiles for quantitative variables. The description will include sociodemographic characteristics (age, sex, years of experience, physical fitness), as well as the analysis of quantitative variables (slope of the relationship between peak velocity and saccadic amplitude, fixation duration in milliseconds, EEG frequency analysis [Theta, Alpha, Beta, Gamma waves], and sleep quantity). Ordinal variables will also be described: Mental Fatigue VAS score, Karolinska Sleepiness Scale (KSS, ordinal 0-9), Morningness-Eveningness Questionnaire (MEQ, ordinal 16-86), Insomnia Severity Index (ISI, ordinal 0-28), and Epworth Sleepiness Scale (ESS, ordinal 0-14).

Analyses for primary and secondary objectives Primary objective

To address the primary objective (assessment of eye movement patterns during a guided saccade task), the investigators will perform a linear regression adjusted for age, years of experience, physical fitness, pre-study fatigue levels, and sleep duration on the day preceding measurement. The independent variable will be the measurement condition (Night shift vs. Rested night), and the dependent variable will be the slope of the relationship between peak velocity and saccadic amplitude during chest X-ray reading.

Secondary objectives Oculomotor behaviour - To evaluate the impact of sleep debt on radiologists' oculomotor behaviour during chest medical image interpretation, the investigators will perform a linear regression adjusted for the same covariates. The dependent variables will be fixation durations (ms) on regions of interest and pupil diameters.

Detection performance - To assess the effect of sleep debt on the number of detected pulmonary embolisms (% detection), the investigators will perform a similar linear regression with % detection as the dependent variable.

EEG-based attentional level - To evaluate the effect of sleep debt on attentional level during observation, measured by portable EEG, the investigators will conduct a regression with EEG frequency bands (Theta, Alpha, Beta, Gamma) as dependent variables.

Subjective perception of sleep and sleepiness - To evaluate the impact of sleep debt on self-reported sleep and sleepiness, the investigators will conduct a regression using subjective measures: Karolinska Sleepiness Scale (KSS), Epworth Sleepiness Scale (ESS), and Mental Fatigue VAS.

Handling of Missing Data Measurement errors In the event of actimeter malfunction or removal for a short period (< 1 hour), data will be considered missing at random. Consequently, the data already collected will be averaged over the total period.

Missing questionnaire data If an item is left unanswered, the calculation of the MEQ, Mental Fatigue VAS, ISI, ESS, or KSS score will be invalidated.

If the data remains missing, the participant will not be included in the regression models involving that variable.

Software used Tobii Pro Lab: eye-tracking Actiware software: actimetry data collection EMOTIV Pro Desktop (local data storage): EEG data collection Matlab (local data storage): actimetry and EEG data analysis R (local data storage): statistical analysis

Expected outcomes

The findings will contribute to:

* A better understanding of the relationships between sleep, oculomotor patterns, attention, and diagnostic performance in radiology.
* Increased awareness of the importance of sleep quality in maintaining optimal analytical performance.
* Evidence to inform organizational changes aimed at minimizing the impact of fatigue, such as adapted shift scheduling or targeted fatigue countermeasures.

This study bridges cognitive neuroscience, medical imaging, and occupational health, with the goal of translating research findings into practical measures to support radiologists' performance and patient safety, particularly in the demanding context of emergency imaging

ELIGIBILITY:
Inclusion Criteria:

Associate radiologists at IMADIS Group

* In their current position for at least one year
* Working at one of the IMADIS Group on-call centers
* Performing night shifts during the study period
* Able to wear an actimeter watch during the study period (it may be removed during certain procedures, but must be put back on afterwards)
* Having given their free and informed consent to participate in the study

Non- inclusion criteria:

* Leave during the study period
* Pregnant women, women in labor, or breastfeeding women
* Subjects wearing glasses or contact lenses

Exclusion Criteria:

- Having slept more than 6 hours during the night shift

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of slope of the relationship between maximum speed and saccade magnitude | Comparison of measurement obtained during an 8-minute guided saccade task during the two measurement phases : after a night call and after a night's rest
  Slope of the relationship between maximum saccadic speed and saccade magnitude This parameter reflects the dynamics of saccadic eye movements. It is derived from the main sequence, which describes the linear relationship between the amplitude of a saccade (in degrees of visual angle) and its maximum velocity (in degrees per second). The slope quantifies how rapidly maximum saccadic speed increases with increasing saccade magnitude. A steeper slope indicates faster oculomotor responses for larger saccades, whereas a reduced slope may reflect fatigue, reduced alertness, or impaired oculomotor function.

SECONDARY OUTCOMES:
Comparison of duration of fixations on areas of interest, in milliseconds | Comparison of measurements taken on the morning after a night shift and on the morning after a night of rest
  Eye tracking measurement performed on pulmonary embolism examination readings. Fixation time measured on areas of interest defined on each examination.
Comparison of percent of embolisms detected | Comparison of measurements taken on the morning after a night shift and on the morning after a night of rest
  Measurement during the reading of chest scans. Information collected using the "logbook" and compared to the gold standard.
Comparison of pupil diameter | Comparison of measurements taken on the morning after a night shift and on the morning after a night of rest
  Pupil diameter measured using eye tracking during the guided saccade task
Comparison of attentional systems | Comparison of measurement taken on the morning after a night shift and on the morning after a night of rest
  EEG measurement of different brain waves (Theta, Alpha, Beta, and Gamma activities) representative of the attentional system.
Assessment of self reported momentary sleepiness | Questionnaire is completed before each measurement phase (after a night on call or after a night of rest)
  using :
  - Karolinska Sleepiness Scale (KSS): is a 9-point self-report measure assessing momentary sleepiness, ranging from 1 = extremely alert to 9 = very sleepy, fighting sleep.
Assessment of self reported habitual daytime sleepiness | Questionnaire is completed before each measurement phase (after a night on call or after a night of rest)
  using : Epworth Sleepiness Scale (ESS) is an 8-item self-report questionnaire evaluating habitual daytime sleepiness in common daily situations, scored from 0-24
Assessment of self reported mental fatigue | Questionnaire is completed before each measurement phase (after a night on call or after a night of rest)
  using : visual analog scale (VAS) for evaluate the mental fatigue (10cm visual scale: 0= no fatigue, 5=medium, 10 extreme)
Assessment of self reported insomnia | Questionnaire is completed before each measurement phase (after a night on call or after a night of rest)
  using : Insomnia Severity Index (ISI) is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia symptoms. Scores range from 0 to 28, with the following thresholds: 0-7 = no clinically significant insomnia, 8-14 = subthreshold insomnia, 15-21 = clinical insomnia of moderate severity, and 22-28 = severe clinical insomnia. A score of 15 or higher will be considered indicative of clinically significant (pathological) insomnia.
Assessment of self reported chronotype | The MEQ questionnaire is completed during inclusion
  using : Morningness-Eveningness Questionnaire (MEQ) is a self-report measure assessing chronotype, determining individual preference for morning or evening activity patterns. Scores range from 16 to 86, with the following thresholds: 16-30 = definite evening type, 31-41 = moderate evening type, 42-58 = intermediate type, 59-69 = moderate morning type, and 70-86 = definite morning type

OTHER OUTCOMES:
Sleep-wake cycle over the last 24 hours | Measurements taken 24 hours before each measurement phase (night shift and a night of rest)
  Measurement taken to determine the subjects' sleep-wake cycle during the 24 hours preceding each measurement. Assessment of the number of hours slept in order to normalize the data during analysis, determined by actimetric measurement

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GORINCOUR, MD, PhD, Principal Investigator — IMADIS Technologies et Services
Locations (1):
- IMADIS Technologies et Services, Lyon, France, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be available upon reasonable request from the principal investigator, after publication of the main results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 2 years after publication.
Access Criteria: Request should be sent by email to the principal investigator, stating the objectives and purpose for using data.
  The request must come from a researcher working in the relevant field of research, and will be reviewed by the scientific committee.
  Principal investigator contact: g.gorincour@imadis-groupe.fr

REFERENCES:
- [Background] Mallett S, Phillips P, Fanshawe TR, Helbren E, Boone D, Gale A, Taylor SA, Manning D, Altman DG, Halligan S. Tracking eye gaze during interpretation of endoluminal three-dimensional CT colonography: visual perception of experienced and inexperienced readers. Radiology. 2014 Dec;273(3):783-92. doi: 10.1148/radiol.14132896. Epub 2014 Jul 15. PMID 25028782
- [Background] Diaz-Piedra C, Rieiro H, Suarez J, Rios-Tejada F, Catena A, Di Stasi LL. Fatigue in the military: towards a fatigue detection test based on the saccadic velocity. Physiol Meas. 2016 Sep;37(9):N62-75. doi: 10.1088/0967-3334/37/9/N62. Epub 2016 Aug 17. PMID 27531394
- [Background] Di Stasi LL, McCamy MB, Macknik SL, Mankin JA, Hooft N, Catena A, Martinez-Conde S. Saccadic eye movement metrics reflect surgical residents' fatigue. Ann Surg. 2014 Apr;259(4):824-9. doi: 10.1097/SLA.0000000000000260. PMID 24169184
- [Background] Gong H, Hsieh SS, Holmes DR 3rd, Cook DA, Inoue A, Bartlett DJ, Baffour F, Takahashi H, Leng S, Yu L, Fletcher JG, McCollough CH. Implementation and initial experience with an interactive eye-tracking system for measuring radiologists' visual search in diagnostic tasks using volumetric CT images. Proc SPIE Int Soc Opt Eng. 2022 Feb-Mar;12031:120310Q. doi: 10.1117/12.2611808. Epub 2022 Apr 4. PMID 35721454
- [Background] De Gennaro L, Ferrara M, Urbani L, Bertini M. Oculomotor impairment after 1 night of total sleep deprivation: a dissociation between measures of speed and accuracy. Clin Neurophysiol. 2000 Oct;111(10):1771-8. doi: 10.1016/s1388-2457(00)00393-x. PMID 11018491
- [Background] Ruutiainen AT, Durand DJ, Scanlon MH, Itri JN. Increased error rates in preliminary reports issued by radiology residents working more than 10 consecutive hours overnight. Acad Radiol. 2013 Mar;20(3):305-11. doi: 10.1016/j.acra.2012.09.028. PMID 23452475
- [Background] Waite S, Kolla S, Jeudy J, Legasto A, Macknik SL, Martinez-Conde S, Krupinski EA, Reede DL. Tired in the Reading Room: The Influence of Fatigue in Radiology. J Am Coll Radiol. 2017 Feb;14(2):191-197. doi: 10.1016/j.jacr.2016.10.009. Epub 2016 Dec 9. PMID 27956140
- [Background] Lee CS, Nagy PG, Weaver SJ, Newman-Toker DE. Cognitive and system factors contributing to diagnostic errors in radiology. AJR Am J Roentgenol. 2013 Sep;201(3):611-7. doi: 10.2214/AJR.12.10375. PMID 23971454
- [Background] West CP, Tan AD, Habermann TM, Sloan JA, Shanafelt TD. Association of resident fatigue and distress with perceived medical errors. JAMA. 2009 Sep 23;302(12):1294-300. doi: 10.1001/jama.2009.1389. PMID 19773564
- [Background] Rollinson DC, Rathlev NK, Moss M, Killiany R, Sassower KC, Auerbach S, Fish SS. The effects of consecutive night shifts on neuropsychological performance of interns in the emergency department: a pilot study. Ann Emerg Med. 2003 Mar;41(3):400-6. doi: 10.1067/mem.2003.77. PMID 12605209
- [Background] Benitez-Provedo C, Talavera B, Garcia-Azorin D, Marcos-Dolado A. The cognitive impact of guard shifts in physicians: a before-after study. Neurol Sci. 2022 Mar;43(3):1701-1708. doi: 10.1007/s10072-021-05501-x. Epub 2021 Aug 18. PMID 34409516
- [Background] Bruls RJM, Kwee RM. Workload for radiologists during on-call hours: dramatic increase in the past 15 years. Insights Imaging. 2020 Nov 23;11(1):121. doi: 10.1186/s13244-020-00925-z. PMID 33226490
- [Background] Bundy JJ, Hage AN, Srinivasa RN, Gemmete JJ, Lee E, Gross JS, Healey TL, Solberg AO, Monroe EJ, Chick JFB. Burnout among Interventional Radiologists. J Vasc Interv Radiol. 2020 Apr;31(4):607-613.e1. doi: 10.1016/j.jvir.2019.06.002. Epub 2019 Jul 22. PMID 31345730